CLINICAL TRIAL: NCT01616420
Title: Assisted Partner Notification to Augment HIV Treatment and Prevention in Kenya
Acronym: APS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Ministry of Health (Other Government); University of Nairobi (Other)
Responsible Party: Principal Investigator, Carey Farquhar, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 43628
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: HIV
Keywords: prevention; treatment; cost-effectiveness; assisted partner notification services; Kenya; linkage to HIV care; case-finding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed aPS (No Intervention)
- Immediate aPS (Experimental)
  Interventions: Other: Assisted-partner notification services

INTERVENTIONS:
Other: Assisted-partner notification services — Assisted-partner notification services (aPS) is a public health service which notifies the partners of those who test positive for a communicable disease of their exposure.
  Other Names: Partner notification services; Assisted partner services
  Arms: Immediate aPS

SUMMARY:
The main purpose of this implementation science study is to find out if providing aPS at 18 different Ministry of Health (MOH) VCT clinics in Kenya works and is cost-effective. This would enable co-investigators in the Kenyan MOH to justify funding to scale-up these services.

The primary aim of the study is to find out whether providing aPS to sexual partners of newly tested HIV-infected individuals can result in more sexual partners getting counseled and HIV tested and linked to HIV care programs for initiation of ART if appropriate. The investigators hypothesize that aPS will increase rates of case-finding, linkages to care, and ART initiation and will not result in social harm.

The second aim is whether aPS is cost-effective in the Kenyan setting. The investigators will estimate how much it costs (when compared to standard methods) to identify and link HIV-infected persons into care. The investigators will also determine how successful aPS is at preventing future HIV transmission events and other outcomes associated with untreated HIV infection. The investigators hypothesize that HIV prevalence among partners in the immediate aPS arm will be high enough to make this approach cost-effective from the payer and societal perspective.

Finally, with the Kenya MOH, the investigators want to establish a nationwide monitoring system to evaluate why Kenyans are testing for HIV. In the future, when aPS is rolled out nationally, this will help Kenyan public health officials define the contribution of aPS to HIV case-finding. The investigators hypothesize that the proportion of newly tested HIV-infected individuals who report testing because of known exposure to a person with HIV will represent a significant proportion of new cases and the investigators will be able to identify places in Kenya where aPS will have the greatest impact on HIV treatment and prevention.

DETAILED DESCRIPTION:
Diagnosing HIV soon after infection can benefit individuals and also has important public health benefits. It has been shown that starting antiretroviral therapy (ART) before HIV has progressed results in a better response to treatment and gives the person a better chance of long-term survival with HIV. Treating HIV can also reduce the risk that someone will transmit HIV to his or her sexual partners. The first step in achieving these individual and population level benefits is testing people for HIV. Unfortunately, in many parts of the world, including Kenya where we plan to conduct this study, many people are not tested regularly and do not know that they are infected. This study involves providing a public health service, notification of an exposure to a communicable disease and HIV testing, to sexual partners of those who test HIV-positive at voluntary counseling and testing (VCT) clinics in Kenya. Sexual partners are identified voluntarily by the person who tests at the VCT. A public health provider then goes to the home of the sexual partners to offer them HIV counseling and testing. This process is called provision of assisted partner services (aPS).

We propose a cluster randomized clinical trial which will be conducted in collaboration with the Kenya Ministry of Health (MOH) at 18 rural and urban voluntary counseling and testing (VCT) facilities across Kenya. Proposed activities will assess the effectiveness and cost-effectiveness of providing aPS, improve capacity for program implementation in Kenya, and lay the foundation for evaluating the program's impact at the national level.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is required of all participants. All participants must be 18 years or older.
* Index case participants must be HIV-seropositive, and willing and able to provide locator information for sexual partners in the past three years.

Exclusion Criteria:

* Index cases will be excluded from participation if they are pregnant, or have reported intimate partner violence during the last month. There is no exclusion criteria for partner participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2424 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of partners testing for HIV | 6 week period following index case enrollment
  The number of partners of an index participant that were tested for HIV (offset will be the number of partners with locator information provided by the index participant).
Newly tested HIV-infected partners | 6 week period following index case enrollment
  The number of partners of an index participant identified as HIV-infected (offset will be the number of partners of that index participant who were HIV tested).
Number of partners linking to HIV care | 6 week period following index case enrollment
  The number of partners of an index participant who were linked to HIV care (offset will be the number of partners of an index participant identified as HIV-infected and analysis will be limited to index participants with at least one HIV-infected partner.)

SECONDARY OUTCOMES:
Incremental cost-effectiveness from payer and societal perspectives | 6 week period following index case enrollment
Proportion of individuals with newly diagnosed HIV infection who report testing because of known exposure to a person with HIV | 6 week period after index case enrollment
Costs of identifying >1 partner per index case | 6 week period after index case enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Carey Farquhar, MD, MPH, Principal Investigator — University of Washington; Peter Cherutich, MBChB, MPH, Study Chair — Kenya Ministry of Health; Matthew Golden, MD, MPH, Study Chair — University of Washington
Locations (18):
- Kenya (18):
  - Karuri VCT, Kiambu
  - Kiambu Hospital VCT, Kiambu
  - Kirwara VCT, Kiambu
  - Chulaimbo Health Centre, Kisumu
  - Joo Trh Vct, Kisumu
  - Kisumu East District Hospital, Kisumu
  - Kombewa VCT, Kisumu
  - Maseno Mission, Maseno
  - Baba Dogo VCT, Nairobi
  - Casino VCT, Nairobi
  - Huruma Lions, Nairobi
  - Kariobangi VCT, Nairobi
  - Kenyatta National Hospital (KNH) VCT, Nairobi
  - Mama Lucy Kibaki VCT, Nairobi
  - Mbagathi VCT, Nairobi
  - Pumwani VCT, Nairobi
  - Abidha Health Centre, Siaya
  - Ongielo Health Centre, Siaya

REFERENCES:
- [Derived] Cherutich P, Golden MR, Wamuti B, Richardson BA, Asbjornsdottir KH, Otieno FA, Ng'ang'a A, Mutiti PM, Macharia P, Sambai B, Dunbar M, Bukusi D, Farquhar C; aPS Study Group. Assisted partner services for HIV in Kenya: a cluster randomised controlled trial. Lancet HIV. 2017 Feb;4(2):e74-e82. doi: 10.1016/S2352-3018(16)30214-4. Epub 2016 Nov 30. PMID 27913227
- [Derived] Wamuti BM, Erdman LK, Cherutich P, Golden M, Dunbar M, Bukusi D, Richardson B, Ng'ang'a A, Barnabas R, Mutiti PM, Macharia P, Jerop M, Otieno FA, Poole D, Farquhar C. Assisted partner notification services to augment HIV testing and linkage to care in Kenya: study protocol for a cluster randomized trial. Implement Sci. 2015 Feb 13;10:23. doi: 10.1186/s13012-015-0212-6. PMID 25884936